CLINICAL TRIAL: NCT02440217
Title: Abnormal Glucose Tolerance is Associated With a Reduced Myocardial Metabolic Flexibility in Patients With Dilated Cardiomyopathy
Brief Title: Myocardial Metabolism in Patients With Dilated Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Associate Professor, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: CardMet
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Dilated Cardiomyopathy; Type 2 Diabetes
MeSH Terms: conditions — Cardiomyopathy, Dilated; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- DCM-AGT: Subjects with both dilated cardiomyopathy (DCM) and abnormal glucose tolerance (AGT, either impaired glucose tolerance or type 2 diabetes).
- DCM-NGT: Subjects with dilated cardiomyopathy (DCM) and normal glucose tolerance (NGT).
- N-AGT: Subjects without dilated cardiomyopathy (N) with abnormal glucose tolerance (AGT, either impaired glucose tolerance or type 2 diabetes).

SUMMARY:
Dilated cardiomyopathy (DCM) is characterized by a metabolic shift from fat to carbohydrates and failure to increase myocardial glucose uptake in response to workload increments. The investigators aimed at verifying whether this pattern is influenced by the presence of abnormal glucose tolerance (AGT).

DETAILED DESCRIPTION:
A catheter is advanced into the coronary sinus by fluoroscopy to withdraw venous blood. A unipolar pacing catheter is positioned into the right atrium. Arterial sampling is done from the femoral artery introducer catheter.

The study protocol consisted of 3 steps (Rest, Pacing and Recovery), during which timed blood samples are collected to measure plasma NEFA and glucose. After the instrumentation is completed, Rest arterio-venous sampling is performed at time -15 min and 0 min. After the 0 min, heart rate is increased by atrial pacing to 110 bpm for 3 minutes and to 130 bpm for 3 additional minutes and arterio-venous sampling is repeated at the end of each step (at time 3 and 6 min). Pacing is then stopped and at time 1, 5, 15 and 30 min into the Recovery period other pairs of arterial and venous samples are withdrawn.

ELIGIBILITY:
Inclusion Criteria:

For patients with dilated cardiomyopathy:

* Myocardial left ventricular ejection fraction (LVEF) <40%
* left ventricular end-diastolic diameter (LVEDD) >56 mm

For patients without dilated cardiomyopathy:

* LVEF >50%
* LVEDD <56 mm.

Exclusion Criteria:

* NYHA class IV
* Atrial fibrillation
* Previous myocardial infarction
* Valvular heart disease
* Myocarditis
* Pericarditis
* Severe to moderate systemic arterial hypertension
* Fasting hyperglycaemia (>7.0 mmol/l)
* Treated diabetes, autoimmune diseases, neoplasia, kidney, liver or respiratory failure

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiology Department of the Institute of Clinical physiology
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial metabolic responses to stress in humans | Arterio-venous sampling will be performed in about an hour during three experimental condition: rest (time -15 and 0 min), pacing (3 and 6 min), and recovery (1, 5, 15 and 30 min).
  The investigators aimed at evaluating myocardial NEFA and glucose uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Professor, Study Chair — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

REFERENCES:
- [Background] Stanley WC, Recchia FA, Lopaschuk GD. Myocardial substrate metabolism in the normal and failing heart. Physiol Rev. 2005 Jul;85(3):1093-129. doi: 10.1152/physrev.00006.2004. PMID 15987803
- [Background] Neglia D, De Caterina A, Marraccini P, Natali A, Ciardetti M, Vecoli C, Gastaldelli A, Ciociaro D, Pellegrini P, Testa R, Menichetti L, L'Abbate A, Stanley WC, Recchia FA. Impaired myocardial metabolic reserve and substrate selection flexibility during stress in patients with idiopathic dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2007 Dec;293(6):H3270-8. doi: 10.1152/ajpheart.00887.2007. Epub 2007 Oct 5. PMID 17921325
- [Derived] Trico D, Baldi S, Frascerra S, Venturi E, Marraccini P, Neglia D, Natali A. Abnormal Glucose Tolerance Is Associated with a Reduced Myocardial Metabolic Flexibility in Patients with Dilated Cardiomyopathy. J Diabetes Res. 2016;2016:3906425. doi: 10.1155/2016/3906425. Epub 2015 Dec 21. PMID 26798650